CLINICAL TRIAL: NCT06200025
Title: The Virtual Reality Rises; The Fall of The Aphasia
Brief Title: Virtual Reality in Aphasia Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Ramazan KURUL, Assistant Professor, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AIBU-FTR-BENLI-006
Record Dates: First submitted 2023-12-29; First posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-12

CONDITIONS: Stroke, Ischemic; Aphasia
MeSH Terms: conditions — Ischemic Stroke; Aphasia

STUDY DESIGN:
Intervention Model Description: two groups with a conventional control group
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Group (Experimental): visual and auditory cue-based aphasia rehabilitation program in full immersive virtual reality
  Interventions: Other: Cue-based speech therapy in virtual reality
- Conventional Group (Active Comparator): visual and auditory cue-based aphasia rehabilitation program
  Interventions: Other: Cue-based speech therapy

INTERVENTIONS:
Other: Cue-based speech therapy in virtual reality — Treatment applied with virtual reality headsets to provide 3d visual and auditory cues to individuals in a virtual environment. A treatment environment where the provision of cues can be controlled by the therapist, interacting with 3d clues and receiving feedback on the accuracy of the named objects.
  Arms: Virtual Reality Group
Other: Cue-based speech therapy — Treatment involving the assessment of language skills and the presentation of communication strategies to the individual, including the use of personalized phonological cues.
  Arms: Conventional Group

SUMMARY:
Virtual reality-based aphasia rehabilitation has been shown to improve the language skills of individuals with aphasia in the chronic period after stroke. However, non-immersive or semi-immersive rehabilitation methods have often been adopted in the studies. Considering the importance of the visual given to the patient for naming, it can be thought that full immersive therapy may be more effective. Therefore, the aim of this study was to investigate the effect of cue-based aphasia naming therapy in a fully immersive virtual reality environment on aphasia severity and aphasia-related quality of life and to compare it with standard cue treatments.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with non-fluent aphasia by a neurologist
* at least 4 months after stroke
* A score of 29 and above on the language score sub-item of the GAT scale

Exclusion Criteria:

* severe sensory impairments (vision, hearing) that prevent participation in therapies
* severe motor dysfunction
* apraxia
* neglect
* dementia
* psychiatric disorders
* 3D vision problems

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Gülhane Aphasia Test | through study completion, an average of 1 year
  Gülhane Aphasia Test-2 (GAT-2) was used to assess aphasia severity. GAT-2 is a valid and reliable test developed by Maviş et al. to evaluate aphasia and to obtain information about motor speech disorders such as dysarthria and apraxia that may accompany aphasia.
  The GAT-2 consists of 7 subsections: speech fluency, listening comprehension, reading comprehension, oral-motor evaluation, automatic speech, repetition and naming. A maximum total score of 82 can be obtained and higher scores are associated with better speech function.

SECONDARY OUTCOMES:
Stroke and Aphasia Quality of Life Scale-39 (SAQOL-39) | through study completion, an average of 1 year
  It is a 39-item valid and reliable scale used to assess quality of life in individuals with aphasia, which examines 4 sub-headings: physical, psychosocial, communication and energy. In 21 items of the scale, the difficulties experienced by individuals with aphasia in their activities in the last week are evaluated, and in the other 18 items, the emotional reactions and possible problems experienced by individuals in the last week are questioned.

CONTACTS AND LOCATIONS:
Overall Officials: Ramazan Kurul, Ph.D, Principal Investigator — Abant Izzet Baysal University
Locations (1):
- Faculty of Health Sciences Bolu Abant Izzet Baysal University, Bolu, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No